CLINICAL TRIAL: NCT03046472
Title: Physical Therapy Treatment Once a Month Versus Physical Treatment Once a Week for Posture Improvement in Children and Adolescents Who Suffer From Posture Problem or Low Back Pain
Brief Title: Physical Therapy Treatment Once a Month Versus Once a Week for Posture Improvement in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Assuta-0133-16-ASMC-AP-CTIL
Record Dates: First submitted 2017-02-05; First posted 2017-02-08 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2017-02

CONDITIONS: Postural Kyphosis, Thoracic Region
Keywords: thorax curve angle
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: The study will consist of two groups: a Treatment group and a control group. Both groups will get personal meeting once a month and a program of exercising at home every day. Treatment group will have in addition group meeting once a week and control group not.
Who Masked: Investigator
Masking Description: One of the investigators has the role of examining the participants before and after the intervention. She will be blinded from the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Once a month and once a week. (Experimental): Personally meeting once a month of Physical Therapy treatment for Postural Behavior.
  In addition exercise group meeting once a week. The intervention program will include physical awareness by using a mirror and practice for good posture, and exercises for flexibility, strength and muscle endurance.
  All participants will get 10-15 minutes of exercise for performing every day. The Participants in this group will get also a group exercise meeting once a week That meeting will long 45 minutes and will include the exercise that were given as home work and more.
  Total duration 12 weeks/3 months
  Interventions: Other: Physical Therapy treatment for Postural Behavior
- Once a month only. (Active Comparator): Personally meeting once a month only for Physical Therapy treatment for Postural Behavior.
  The intervention program will include physical awareness by using a mirror and practice for good posture, and exercises for flexibility, strength and muscle endurance.
  All participants will get 10-15 minutes of exercise for performing every day. Total duration 12 weeks/3 months
  Interventions: Other: Physical Therapy treatment for Postural Behavior

INTERVENTIONS:
Other: Physical Therapy treatment for Postural Behavior — Physical Therapy treatment for Postural Behavior: intervention program will include physical awareness by using a mirror and practice for good posture, and exercises for flexibility, strength and muscle endurance.
  All participants will get 10-15 minutes of exercise for performing every day.

SUMMARY:
This study is design in a clinical setting for testing whether physical therapy treatment that includes postural awareness exercises for strength flexibility and endurance is improving low back pain and postural behavior. The study will consist of two groups, basic treatment that will get one on one treatment once a month for 3 months and the intervention group, will get an additional group therapy once a week.

DETAILED DESCRIPTION:
Background: Life time prevalence of Low Back Pain among Children and Adolescent ranges from 32% to 66%. This prevalence gets higher with age and among 17 years old it's equal to prevalence among adults. Previous episode of Low Back pain is a predicting risk factor to the next one, hence we should do preventative care at a young age, even before the first attack occur. Poor posture was found as one of the risk factors for Low Back Pain in children. Adolescence with neutral posture had less prevalence of Low Back Pain then those with poor posture. Prolong slouch sitting was associated with Low Back Pain. Prevention education programs, focusing on knowledge, did not show effective change in posture behavior. Hence, the researchers concluded that it's better if they focus on exercise.

Research Goal: comparison between physical therapy treatment for good posture once a week versus once a month, on postural behavior, thorax curve angle and Low Back Pain.

Research type: randomize, Interventional, blinded. Methods and Procedures Population: the study will include 50 children and adolescents age 10-18 years suffering from poor back posture, with or without Low Back Pain.

Procedure: The study will consist of two groups: both groups will get personal meeting once a month and a program of exercising at home every day. Treatment group will have in addition group meeting once a week and control group not. The intervention program will include physical awareness and practice for good posture, and exercises for flexibility, strength and muscle endurance.

Measurement tools:Digital Inclinometer for measuring thorax curve angle. Postural observation for measuring postural habits. Back pain and postural habits questionnaire for measuring LBP on VAS SCALE, postural knowledge and habits of participant, including demographic data. Parents' questionnaire for measuring parents' knowledge and ideas.

Research hypothesis: postural behavior, thorax curve angle and Low Back Pain will get better in both groups but more in the treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Children and Adolescent who referred by their pediatrician or orthopedic doctor to Physical Therapy treatment due to bad posture or Low Back Pain
2. At the Physical Therapy clinic was found that this is truly the condition of bad posture or low back pain with bad posture.
3. age 10-18 years
4. they signed on informed consent.

Exclusion Criteria:

1. Children and Adolescent who suffer from risk of structural deterioration as structural scoliosis(Cob angle above 20° and Risser sign equal or below 3) or structural Kyphosis (above 40° Risser sign equal or below 3 or Scheuermann Disease)
2. Any sever health condition neurologic internal or orthopedic like Cerebral Palsy, Juvenile rheumatoid arthritis or Malignancy.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asaf Peretz, MD, Principal Investigator — Deputy Medical Director-Maccabi Health Services-Jerusalem hashfela; Neta Vitman, PT BA, Study Director — Phisical Therapy Maccabi Health services-Modiin Clinic
Locations (1):
- Phisical Therapy Clinic Maccabi Health Services, Modiin, Jerusalem-Hashfela, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Once a Month Only.: Personally meeting once a month only for Physical Therapy treatment for Postural Behavior.
  The intervention program will include physical awareness by using a mirror and practice for good posture, and exercises for flexibility, strength and muscle endurance.
  All participants will get 10-15 minutes of exercise for performing every day. Total duration 12 weeks/3 months
  Physical Therapy treatment for Postural Behavior: Physical Therapy treatment for Postural Behavior: intervention program will include physical awareness by using a mirror and practice for good posture, and exercises for flexibility, strength and muscle endurance.
  All participants will get 10-15 minutes of exercise for performing every day.
- Once a Month and Once a Week.: Personally meeting once a month of Physical Therapy treatment for Postural Behavior.
  In addition exercise group meeting once a week. The intervention program will include physical awareness by using a mirror and practice for good posture, and exercises for flexibility, strength and muscle endurance.
  All participants will get 10-15 minutes of exercise for performing every day. The Participants in this group will get also a group exercise meeting once a week That meeting will long 45 minutes and will include the exercise that were given as home work and more.
  Total duration 12 weeks/3 months
  Physical Therapy treatment for Postural Behavior: Physical Therapy treatment for Postural Behavior: intervention program will include physical awareness by using a mirror and practice for good posture, and exercises for flexibility, strength and muscle endurance.
  All participants will get 10-15 minutes of exercise for performing every day.
Period: Overall Study
Arm/Group | Once a Month Only. | Once a Month and Once a Week.
Started | 33 | 17
Completed | 33 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Once a Month and Once a Week. | Once a Month Only. | Total
Number analyzed (Participants) | 17 | 33 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 33 | 50
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.2 (2.1) | 14.0 (1.9) | 14.2 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 16 | 26
  Male | 7 | 17 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Israel | 17 | 33 | 50
Thorax curve angel [Mean (Standard Deviation); unit: degrees] | 39.2 (9.3) | 38.9 (9.3) | 39.0 (9.8)
Low back Pain in VAS Scale [Mean (Standard Deviation); unit: units on scale 0-10] — we asked the patient if they suffered from back pain in period of 3 months previous that day on Vas scale 0-10 0 no pain 1-2 very mild pain 2-3 mild pain 4-6 moderate pain 7-8 high pain 9-10 very high pain Population: not all participants had Low Back Pain
  units on scale 0-10
    number analyzed (Participants) | 12 | 21 | 33
    (all) | 5.6 (2.2) | 5.5 (2.1) | 5.5 (2.1)
Overall Back Postural Behavior [Mean (Standard Deviation); unit: units on scale 0-16] — Overall postural behavior: The patient observation was comprised of 8 observations including: waiting for treatment, walking into the room, sitting, laying mattress on the floor, exercises on four pose, sitting and standing poses, and the transition between them. Each observation was graded as 0=poor, 1=fair, 2=good, summarized into grades 0 to 16.An higher score is a better behavior.
  units on scale 0-16 | 2.1 (1.8) | 2.2 (2.4) | 2.2 (2.2)
spontaneous Back Postural Behavior [Mean (Standard Deviation); unit: units on scale 0-8] — Spontaneous behavior was defined as the summation of four of the overall observations who has a spontaneous characteristics : waiting for treatment, walking into the room, sitting in treatment and transition between poses, each of them was graded as 0=poor, 1=fair, 2=good, summarized into grades 0-8.
  An higher score indicates a better behavior.
  units on scale 0-8 | 0.5 (0.8) | 0.5 (0.9) | 0.5 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Thoracic Kyphosis Angle
Description: Normal thoracic kyphosis angle ranges between 25°-40°. Measuring by Digital Inclinometer by placing it on the spinous process of T1 and T12 and the outcome off subtraction the two numbers is our out come.
  The participant is to stand how ever he think is the best posture.
Time Frame: 2 time points. before starting intervention and after 3 months.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Once a Month Only. | Once a Month and Once a Week.
Number analyzed (Participants) | 33 | 17
degrees
  Curve angle baseline | 39.2 (9.3) | 38.9 (9.3)
  Curve angle end | 27.9 (7.8) | 28.2 (6.8)
Statistical Analysis 1: Comparison: Once a Month Only. vs Once a Month and Once a Week; Test type: Other; p < 0.001, ANOVA

2. Primary Outcome: Low Back Pain
Description: VAS Scale 0-10 0 no pain 1-2 very mild pain 2-3 mild pain 4-6 moderate pain 7-8 high pain 9-10 very high pain
Time Frame: 2 time points. before starting intervention and after 3 months.
Population: only 33 out of 50 had LBP 21 in once a month group and 12 in once a month and once a week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Once a Month Only. | Once a Month and Once a Week.
Number analyzed (Participants) | 21 | 12
score on a scale
  LBP Baseline | 5.5 (2.1) | 5.6 (2.2)
  LBP End | 2.8 (2.0) | 1.6 (1.9)
Statistical Analysis 1: Comparison: Once a Month Only. vs Once a Month and Once a Week; Test type: Other; p < 0.001, ANOVA

3. Primary Outcome: Back Postural Behavior
Description: the investigator observes the participant in 8 different positions: sitting in the waiting room, walking to the treatment room, sitting in front of the therapist, placing a mattress on the floor, exercising in six position, exercising in sitting position, exercising in standing position, and changing between positions. Each position get a subscore as 0-bad posture 1-fair 2-good. Overall postural behavior: was comprised of all 8 observations including: grades 0 to 16. An higher score is a better behavior.
  spontaneous behavior was comprised of 4 sob score that ha a spontaneous characteristics: sitting waiting for treatment, walking into the room, sitting during treatment and transition between exercises. summation of these 4 would range 0-8 . an Higher score is a better behavior.
Time Frame: 2 time points. before starting intervention and after 3 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Once a Month Only. | Once a Month and Once a Week.
Number analyzed (Participants) | 33 | 17
score on a scale
  Difference Overall back postural behavior | 6.7 (3.1) | 9.0 (2.3)
  Difference spontaneous back postural behavior end | 3.0 (1.9) | 4.1 (1.7)
Statistical Analysis 1: Comparison: Once a Month Only. vs Once a Month and Once a Week; Test type: Other; p = 0.01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 months for each patient. total time of collecting data no more then 10 months
Arm/Group | Once a Month Only. | Once a Month and Once a Week.
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/17
Other Adverse Events (participants affected / at risk) | 0/33 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/72/NCT03046472/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/72/NCT03046472/SAP_001.pdf